CLINICAL TRIAL: NCT07219134
Title: Pilot Investigation of Dual Energy CT Imaging on an Online Adaptive Radiation Therapy System
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Varian Medical Systems, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: UMCC 2024.027; NCI-2025-03767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00259510 (Other: University of Michigan)
Record Dates: First submitted 2025-08-11; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Genitourinary System Carcinoma; Malignant Pelvic Neoplasm
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational: Patients undergo lower beam energy CBCT scan once during standard of care radiation therapy on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to see if researchers can find a better way to image a patient's tumor during radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* * Patients with pelvis or genitourinary (GU) cancer requiring standard of care radiotherapy treatment

  * All adults, defined as individuals of 18 years of age or greater
  * Radiotherapy treatment will be performed on the Varian Ethos radiotherapy system
  * Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* * Minors, defined as individuals less than 18 years of age

  * Pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pelvis or genitourinary cancer requiring standard of care radiotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Image quality- Mean | Up to 2 years
  The primary analysis will compare imaging quality endpoints processed by DE-CBCT and the standard of care SE-CBCT, with the latter representing the standard clinical acquisition. Descriptive statistics will be computed for the image quality metrics from each imaging modality and for the difference in metrics between the modalities. A paired t-test or Wilcoxon signed-rank test will compare the distribution of the image quality metrics between DE-CBCT and standard of care SE-CBCT. Secondary analysis will compare image quality endpoints between DE-CBCT and standard of care conventional planning CT.
Image quality- median | Up to 2 years
  The primary analysis will compare imaging quality endpoints processed by DE-CBCT and the standard of care SE-CBCT, with the latter representing the standard clinical acquisition. Descriptive statistics will be computed for the image quality metrics from each imaging modality and for the difference in metrics between the modalities. A paired t-test or Wilcoxon signed-rank test will compare the distribution of the image quality metrics between DE-CBCT and standard of care SE-CBCT. Secondary analysis will compare image quality endpoints between DE-CBCT and standard of care conventional planning CT.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dess, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No